CLINICAL TRIAL: NCT01759940
Title: Influence of the Concentration of the Local Anesthetic Ropivacaine on the Quality of a Ultrasound Guided Block of the Regio Collis Lateralis for Carotid Endarterectomy: a Prospective, Randomized and Controlled Trail
Brief Title: Influence of the Concentration of the Local Anesthetic Ropivacaine on the Quality of a Ultrasound Guided Intermediate Cervical Block.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Andreas Kokoefer, MD, Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cervicalblock; 2012-002769-37 (EudraCT Number)
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Intermediate Cervical Plexus Block for Carotid Endarterectomy
Keywords: carotid; endarterectomy; cervical block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine 0,375% (Experimental): In the study group the intermediate cervical block will be performed by ultrasound guidance using 20ml ropivacaine 0,375%. Additionally 10ml prilocaine 1% will be used to infiltrate the perivascular tissue around the carotid artery. In the area of the expected incision the skin will also be infiltrated with 10ml prilocaine 1%.
  Interventions: Drug: ropivacaine 0,375%
- ropivacaine 0,75% (Active Comparator): In the control group the intermediate cervical block will be performed by ultrasound guidance using 20ml ropivacaine 0,75%. Additionally 10ml prilocaine 1% will be used to infiltrate the perivascular tissue around the carotid artery. In the area of the expected incision the skin will also be infiltrated with 10ml prilocaine 1%.
  Interventions: Drug: ropivacaine 0,75%

INTERVENTIONS:
Drug: ropivacaine 0,375%
  Arms: ropivacaine 0,375%
Drug: ropivacaine 0,75%
  Arms: ropivacaine 0,75%

SUMMARY:
Carotid endarterectomy is commonly performed under cervical plexus block. This is presumed to offer advantages over general anesthesia in terms of monitoring neurological function during cross-clamping of the carotid artery since, in conscious patients, speech, cerebration, and motor power provide early measures of inadequate cerebral perfusion. Some studies also claim lower shunting requirements, lower cardiovascular morbidity, and shorter hospital stay.

Traditionally, the common methods of cervical plexus block are termed 'deep' or 'superficial'. The deep block, as described by Moore or Winnie and colleagues, consists of identifying the transverse processes of upper cervical vertebrae C2 - C4 and injecting local anesthetic directly into the deep (prevertebral) cervical space. This may be achieved either as separate injections or as a single injection. The superficial block incorporates a variety of procedures. The simplest is a s.c. infiltration of local anesthetic along the posterior border of sternocleidomastoid muscle by either the surgeon or the anesthetist.

An 'intermediate' block is one where the injecting needle pierces the investing fascia of the neck, deep to the s.c. layer, but superficial to the deep cervical (prevertebral) fascia. It is also possible to use a 'combined block', consisting of a deep injection and a superficial or intermediate injection.

Practitioners may prefer one block to another, but no consensus exists on the efficacy of one block when compared with another. However, it has been suggested that complications of the technique are related to the deep injection and not the superficial (or intermediate) injection. These complications include intrathecal or intravascular injection, respiratory problems related to phrenic nerve paralysis, or local anaesthetic toxicity.

In this study the Influence of the concentration of the local anesthetic ropivacaine on the quality of the intermediate cervical plexus block for carotid endarterectomy will be evaluated. For this purpose two different concentrations of ropivacaine will be compared (3,75% vs 7,5%). The primary endpoint of the study will be the quantity of the additional needed local anesthetic to achieve adequate operative analgesia. Furthermore we will record the frequency of the most common side effects as well as the patient satisfaction with a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for carotid endarterectomy in regional anesthesia

Exclusion Criteria:

* refusal to participate in the trail
* age < 18a
* gestation/breastfeeding
* contraindication for regional anesthesia
* inclusion in other trails

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
amount of additional needed local anesthetics by the surgeon | The primary endpoint will be evaluated continuously during the ongoing surgery by interrogating the patients pain scale every two to five minutes. In average the whole procedure will take 30 to 50 minutes.
  The surgeon will titrate the local anesthetic lidocaine 2%to achieve adequate operative analgesia for the patient. During the surgical procedure the patient will not be sedated therefore distinct communication to the patient is always possible.

SECONDARY OUTCOMES:
plasma concentrations of ropivacaine | until 8h postoperative
  measured with mass spectrometry
vital signs | whole day of surgery
  continuous recording of vital signs during the surgery as well as in the postoperative ICU
effect on the diaphragm function | until 6 h postoperative
  assessment of phrenic nerve paresis by ultrasound measurement of the diaphragm excursions, performed by the radiologist on call

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kokoefer, MD, Principal Investigator — Salk Institute for Biological Studies
Locations (1):
- Klinik für Anästhesiologie, perioperative Medizin und allgemeine Intensivmedizin, Salzburg, Salzburg, Austria

REFERENCES:
- [Derived] Kokofer A, Nawratil J, Felder TK, Stundner O, Mader N, Gerner P. Ropivacaine 0.375% vs. 0.75% with prilocaine for intermediate cervical plexus block for carotid endarterectomy: A randomised trial. Eur J Anaesthesiol. 2015 Nov;32(11):781-9. doi: 10.1097/EJA.0000000000000243. PMID 25782662